CLINICAL TRIAL: NCT06350383
Title: Adapting a Low-cost Intimate Partner Violence (IPV) and Mental Health Response Intervention for Women in Informal Settlements in Kenya
Brief Title: Adapting a Low-cost Intimate Partner Violence and Mental Health Response Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Drexel University (Other); Africa Mental Health Research and Training Foundation (Unknown); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Samantha C. Winter, Associate Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AAAT8527; K01TW011775 (NIH)
Record Dates: First submitted 2024-03-14; First posted 2024-04-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Violence, Domestic; Psychological Distress
Keywords: Intimate partner violence (IPV); Randomized control trial (RCT); Wings of Hope (WINGS); Problem Management Plus (PM+); Kenya; Informal settlements (slums); Women

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group design
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be told to which arm they have been randomized. Additionally, to reduce contamination, community health volunteers (CHVs) will either carry out assessment or intervention, not both. Assessors will not be told to which arm participants they are assessing have been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WINGS+PM+ (Experimental): WINGS+PM+ is a safety, harm reduction, and brief psychological intervention that involves seven 90-minute weekly sessions focused on exploring types and mechanisms of IPV; building motivation to address IPV; safety planning and revision; enhancing social support to address IPV; goal setting and revision; identifying IPV-related services and needs; linkage and referral to services; self-care planning; learning and practicing a stress management technique; identifying, defining, and managing problems through goal setting and review; increasing engagement in positive activities; strengthening social supports; and developing plans to stay healthy and well beyond the intervention.
  Interventions: Behavioral: WINGS+PM+
- PM+-Only (Active Comparator): PM+: is a brief psychological intervention also designed to be facilitated by non-specialists (e.g. CHVs) and focused on problem management and evidence-based behavioral strategies to enhance one's capacity to adaptively manage psychological distress. It has been shown to be effective at reducing psychological distress among women who have experienced gender-based violence in informal settlements in Nairobi, Kenya. PM+ involves five 90-minute, weekly individual sessions focused on learning and practicing a stress management technique; identifying, defining, and managing problems through goal setting and review; increasing engagement in positive activities; strengthening social supports; and developing plans to stay healthy and well beyond the intervention.
  Interventions: Behavioral: PM+-only

INTERVENTIONS:
Behavioral: WINGS+PM+ — WINGS+PM+ is a safety, harm reduction, and brief psychological intervention combined and adapted by community members from informal settlements in Kenya (IPV survivors, health clinic staff, and CHVs) from two evidence-based interventions: Wings of Hope (WINGS) and Problem Management Plus (PM+). This intervention was designed to be facilitated by non-specialists (e.g., CHVs). It involves seven 90-minute weekly sessions. The intervention is informed by social cognitive theory.
  Arms: WINGS+PM+
Behavioral: PM+-only — PM+: is a brief psychological intervention also designed to be facilitated by non-specialists (e.g. CHVs) and focused on problem management and evidence-based behavioral strategies to enhance one's capacity to adaptively manage psychological distress. It has been shown to be effective at reducing psychological distress among women who have experienced gender-based violence in informal settlements in Nairobi, Kenya. PM+ involves five 90-minute, weekly individual sessions.
  Arms: PM+-Only

SUMMARY:
The goal of this feasibility study (clinical trial) is to test a low-cost, combined, adapted intimate partner violence (IPV) and mental health intervention (Wings of Hope: WINGS + Problem Management Plus: PM+) that can be carried out by lay community health workers as a foundation for a potential low-cost essential services package for women experiencing IPV and related mental health challenges in informal settlements in Kenya. The main aims of the study are to (1) assess the safety, feasibility, and acceptability of WINGS+PM+ among women experiencing IPV in informal settlements in Kenya; (2) to test preliminary efficacy of program mediating outcomes in addition to the distal outcome (incidence/severity of IPV), while closely monitoring fidelity or process measures, including attendance/retention, adherence, quality of delivery, participant satisfaction, safety and quality improvement and adaptation modifications; and (3) generate data on distributions of study outcomes to calculate the power to detect a meaningful effect size in a future efficacy trial. Women experiencing IPV (n=260) will be recruited from the outpatient walk-in departments at the Kianda 42 Hospital in Kibera informal settlement (n=130) and Upendo Clinic in Mathare informal settlement (n=130). Consenting women will be screened for experiences of recent IPV (last 3 months). Subsequently 130 eligible IPV survivors from the Kianda 42 Hospital and 130 from the Upendo Clinic will be randomized to either receive the combined WINGS+PM+ intervention (n=65) or the PM+-only intervention (control/comparison arm) (n=65) at each clinic.

DETAILED DESCRIPTION:
Women experiencing IPV (n=260) will be recruited from the outpatient walk-in departments at Kianda 42 Clinic in Kibera informal settlement (n=130) and Upendo Clinic in Mathare informal settlement (n=130). Consenting patients will be screened for recent experiences of IPV (past 3 months) by nurses or staff using an adapted version of the World Health Organization (WHO) IPV Brief Self-screener (IPV-BSS) and asked several mental health and functioning questions.

Informational scripts about the study will be shared and posted at the two clinics and also shared by community health volunteers (CHVs) with clinic patients during routine household visits. Every CHV who is attached to a clinic is responsible for doing routine visits with clinic patients in up to 100 households each month in the informal settlement in which the clinic is located. The purpose of these routine household visits is to check-in on patients, let households know about new or relevant clinic programs, and carry out relevant health-related trainings (e.g., how to treat water during a cholera outbreak or how to practice proper hygiene during COVID). The informational script will let patients in the clinics and broader community know that, if they are interested in the program, they can come to the clinic to be screened for eligibility.

Eligibility/IPV screens will be collected by trained non-specialist in-take staff in a private in-take room at the Kianda 42 Clinic in Kibera and Upendo in Mathare. Screening is anonymous. No identifying information will be collected as part of the screen. Answers to the screening questions will be recorded on digitally on study tablets. Verbal consent for eligibility screens will be collected. In-take staff will note on the informed consent document that the participant verbally consented to the screening, and sign their own names to attest to participants' consent.

If women screen positive for IPV in the past three months and meet the rest of the eligibility criteria, they will be asked if they are interested in participating in the feasibility trial. If they express interest, they will be referred to a trained CHV who will take them through the a digital Informed Consent Process for the feasibility trial.

Consenting participants will be guided through a baseline assessment by a CHV and then randomized to either the combined WINGS+PM+ (n=130; 65 at Kianda 42 and 65 at Upendo) or the psychological-only (PM+) arm (n=130; 65 at Kianda 42 and 65 at Upendo). Block randomization with random block sizes will be used to "force" a balance between study arms with respect to the number of women per arm per clinic.

WINGS+PM+ and PM+-only sessions will be delivered by trained CHVs at Kianda 42 and Upendo. WINGS+PM+ is a safety, harm reduction, and brief psychological intervention combined and adapted by community members from informal settlements in Kenya (IPV survivors, health clinic staff, and CHVs) from two evidence-based interventions: Wings of Hope (WINGS) and Problem Management Plus (PM+). This intervention was designed to be facilitated by non-specialists (e.g., CHVs). It involves seven 90-minute weekly sessions focused on exploring types and mechanisms of IPV (e.g., the role of household economics in IPV); building motivation to address IPV; safety planning and revision; enhancing social support to address IPV; goal setting and revision; identifying IPV-related services and needs; linkage and referral to services; self-care planning; learning and practicing a stress management technique; identifying, defining, and managing problems through goal setting and review; increasing engagement in positive activities; strengthening social supports; and developing plans to stay healthy and well beyond the intervention. PM+: is a brief psychological intervention also designed to be facilitated by non-specialists (e.g. CHVs) and focused on problem management and evidence-based behavioral strategies to enhance one's capacity to adaptively manage psychological distress. It has been shown to be effective at reducing psychological distress among women who have experienced gender-based violence in informal settlements in Nairobi, Kenya. PM+ involves five 90-minute, weekly individual sessions focused on learning and practicing a stress management technique; identifying, defining, and managing problems through goal setting and review; increasing engagement in positive activities; strengthening social supports; and developing plans to stay healthy and well beyond the intervention.

Intervention outcomes will be assessed at four time points: baseline, immediately post intervention (IPI), 3-month, and 6-month follow-up.

To reduce contamination, CHVs will either carry out assessment or facilitate the intervention. Some CHVs will deliver PM+-only while others will deliver the WINGS+PM+ intervention. Project staff will meet regularly with CHVs providing PM+ only to establish the types of support and counselling they offered to participants and check that there was no contamination of the WINGS+PM+ strategies in the PM+-only arm. All intervention sessions will be audio-recorded for quality assurance.

ELIGIBILITY:
Inclusion Criteria:

* Reports experiencing IPV in the past 3 months using the WHO IPV-BSS screener
* Reports feeling safe participating in the study
* Able to provide informed consent and follow study procedures
* Fluent in English and/or Swahili
* At least 18 years of age

Exclusion Criteria:

* Does not report IPV in the past 3 months,
* Does not feel safe participating in study,
* Unable to provide informed consent and/or follow study procedures,
* Cannot communicate in English or Swahili,
* Under the age of 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who self-identify as women are eligible to participate. Sex-at-birth will not be assessed.
Enrollment: 260 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
World Health Organization (WHO) Violence Against Women (VAW) diagnostic instrument | Baseline, immediately post intervention, 3-month follow-up, 6-month follow-up
  A modified version of the WHO-VAW Corr 5 will be used to measure recent experience of IPV. The WHO IPV diagnostic tool has been used in Kenya previously. It includes four subscales measuring controlling behaviors (7 items) and sexual (3 items), physical (6 items), and emotional IPV (4 items). Participants will be asked whether or not (0=no, 1=yes) and the number of times they experienced any of these IPV items in the prior 90 days at baseline, IPI, and the 3- and 6- month follow-up.

SECONDARY OUTCOMES:
Receipt of violence services | Baseline, immediately post intervention, 3-month follow-up, 6-month follow-up
  Receipt of violence-related services will be measured with an item used in prior assessments of WINGS that asks, 'Have you received any services, counselling or group support for partner abuse or violence from others in the past 90 days?'
Domestic Violence Coping Self-efficacy Scale (DVCSE) | Baseline, immediately post intervention, 3-month follow-up, 6-month follow-up
  IPV self-efficacy will be assessed using the DVCSE, a 30-item scale that measures perceived competency in managing abuse and conflict with partners. The items are rated on a 5-point Likert scale ranging from "not at all confident" to "very confident".
Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline, immediately post intervention, 3-month follow-up, 6-month follow-up
  Social Support will be measured with the 12-item MSPSS, which assesses the availability of emotional and instrumental support and advice for relationship conflict or problems with intimate partners and other issues. Items are measured on a 7-point Likert scale ranging from very strongly disagree (1) to very strongly agree. High scores on the scale suggest higher levels of social support.
Safety Behavior Checklist | Baseline, immediately post intervention, 3-month follow-up, 6-month follow-up
  Safety behaviors will be assessed using an updated version of a 7-item safety behavior checklist to determine present use of safety behaviors and to chart future adoption. The adjusted total score falls within a 0-7 range of behaviors performed, with higher scores suggesting more safety behaviors.
Psychological distress (GHQ-12) | Baseline, immediately post intervention, 3-month follow-up, 6-month follow-up
  Psychological distress will be measured with the Kiswahili version of the GHQ-12, which indexes psychological distress, including anxiety and depression, in the past few weeks. The GHQ-12 comprises 12 questions scored on a 4-point scale ranging from 0 to 3 (range 0-36; higher scores indicate more severe psychological distress). A cutoff of 12/13 (using the 4-point continuous scoring system can be used to detect psychological morbidity, as has previously been used in Kenyan trials of the PM+ intervention.
Functioning (WHODAS 2.0) | Baseline, immediately post intervention, 3-month follow-up, 6-month follow-up
  Functional impairment will be measured using the WHODAS 2.0. This 12-item instrument assesses difficulty in completing activities in the last 30 days (range 0-48; higher scores indicate greater impairment severity). The WHODAS 2.0 has been used widely as a screening and outcome measure, demonstrates moderate to strong evidence of construct- and criterion-related validity, displays good sensitivity to change and has been used previously in PM+ efficacy trials in Kenya and in informal settlements in Kenya.
Short form of the Posttraumatic Stress Disorder Checklist (PCL-5) | Baseline, immediately post intervention, 3-month follow-up, 6-month follow-up
  A four-item, short version of the Posttraumatic Stress Disorder Checklist (PCL) will be used to measure symptoms of PTSD. The PCL was adapted and used for an efficacy trial of PM+ in Kenya. Items are scored with a 5-point Likert ranging from 0= "not at all" to 4="extremely", with high scores suggesting symptoms of PTSD.
Personalized outcomes (PSYCHLOPS) | Baseline, immediately post intervention, 3-month follow-up, 6-month follow-up
  The Psychological Outcome Profiles (PSYCHLOPS) scale will be used to assess change in relation to problems that are identified by the participant. It asks respondents to nominate 2 of their main problems and to provide ratings on the magnitude of the problems and their effects on functioning and well-being in the previous week. It is sensitive to change and is internally reliable. PSYCHLOPS assesses the impact of interventions on problems that are not necessarily assessed by other standardized measures; thus, it can be useful in the context of informal settlements, where people can suffer a diverse range of problems. It has also been used in an efficacy trial of PM+ in Kenya.

OTHER OUTCOMES:
Quality control/intervention fidelity | Through study completion, an average of 8 months
  Using monitoring systems from previous studies (adherence to activities and delivery quality checklists), investigators will assess intervention protocol fidelity. Investigators will audiotape all intervention sessions and randomly select and review 15% in order to assess quality control and implementation fidelity. Fidelity levels below 80% will trigger retraining and closer supervision.
Facilitator Satisfaction and ease of intervention delivery (EBPAS-36) | Through study completion, an average of 8 months
  Facilitator satisfaction and ease of intervention delivery will be assessed with a shortened version of the Evidence-Based Practice Attitude Scale (EBPAS-36). Responses are given on a 5-point Likert scale ranging from 0="not at all" to 4="to a very great extent." With high scores indicating satisfaction.
Adverse events | Through study completion, an average of 8 months
  Safety will be assessed through adverse event reporting by CHVs/Research Assistant (RA)/clinic staff and exit interviews with CHVs asking about negative intervention experiences.
Participant satisfaction with intervention | Through study completion, an average of 8 months
  Participants will be asked to rate their satisfaction with the session at the end of each intervention session.
Number of participants in attendance at sessions | Through study completion, an average of 8 months
  Attendance for each participant at each session will be tracked.
Retention Rate | Baseline, immediately post intervention, 3-month follow-up, 6-month follow-up
  Retention through assessment completion will be tracked and, to the extent possible, investigators will follow-up with participants who dropped out to inquire after the reasons for drop out.

CONTACTS AND LOCATIONS:
Locations (2):
- Kenya (2):
  - Upendo Clinic, Nairobi
  - Kianda 42 Hospital, Nairobi

IPD SHARING:
Plan to Share IPD: No